CLINICAL TRIAL: NCT03617783
Title: Prebiotic Treatment in People With Schizophrenia
Brief Title: Prebiotic Treatment in People With Schizophrenia - Pilot Study
Acronym: preFOCIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Robert Buchanan, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HP-00081820
Record Dates: First submitted 2018-07-16; First posted 2018-08-06 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prebiotin (Active Comparator)
  Interventions: Drug: Prebiotin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prebiotin — Prebiotin (12g/day), an oligofructose-enriched inulin (OEI)
  Arms: Prebiotin
Drug: Placebo — placebo-OEI
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine changes in serum butyrate levels with the prebiotic: Prebiotin (12g/day), an oligofructose-enriched inulin (OEI); the effect of OEI on the composition of the gastrointestinal microbiota in people with schizophrenia; and the relationship of the composition of the gut microbiota to various clinical, cognitive, and neuroimaging variables.

DETAILED DESCRIPTION:
Over the past 10 years, considerable evidence has emerged from animal studies to suggest that the gut microbiome has significant effects on brain development and behavior, with bidirectional communication between the enteric nervous system, gut and the central nervous system (CNS) (Diaz Heijtz et al, 2011; Douglas-Escobar et al, 2013; Dinan et al, 2014). The gut microbiota have been shown to: a) produce multiple neurotransmitters, including gamma-aminobutyric acid (GABA), dopamine, norepinepherine, and serotonin, and may regulate CNS levels of these neurotransmitters; b) modulate brain development through the regulation of synaptogenesis; and c) modulate the levels of stress hormones during brain development, which may affect stress response and anxiety behavior (Diaz Heijtz et al, 2011; Dinan et al, 2014; Sudo et al, 2004; O'Mahony et al, 2015). Moreover, the gut microbiota effects the production of neurotrophins, including brain-derived neurotrophic factor (BDNF), which plays a significant role in neurogenesis and synaptic plasticity (Sudo et al, 2004; Nemani et al, 2015).

The gut microbiome may also affect brain development and function through its regulation of immune system function, which is mediated, in part, through the production of short-chain fatty acids (SCFA). There are three major SCFAs: butyrate, propionate, and acetate. Butyrate is of particular interest, since it plays a key role in maintaining gut homeostasis and epithelial integrity: butyrate is the primary energy source for intestinal colonocytes; and, of the three SCFAs, butyrate appears to have the most pronounced effects on immune system function and may exert its effects directly through immune pathways and indirectly through the maintenance of the integrity of the intestinal-blood barrier (Hamer et al, 2008; Louis et al, 2010; Brahe et al, 2013; Vital et al, 2014). The intestinal-blood barrier restricts the entrance of toxins, pathogens and antigens into the blood circulation; thus, increased permeability could lead to the entrance of substances and subsequent immune response.

The multiple effects of the gut microbiome on brain development and behavior, suggest that alterations in the gut microbiome may occur in schizophrenia and play a part in the pathophysiology of the disorder. The increased prevalence of gastrointestinal disorders in schizophrenia; the association of infections, including infections with Toxoplasma gondii, which can induce intestinal inflammation, with the risk for the development of schizophrenia; and evidence of increased gut permeability provide further indirect evidence for disruption of the gut microbiome in this disorder (Dinan et al, 2014; Nemani et al, 2015; Severance et al, 2012; Severance et al, 2014). Although a number of studies have been conducted in other neuropsychiatric disorders, including autism (Parracho et al, 2005; Tomova et al, 2015), which demonstrate altered bacterial composition of the gut microbiome, there is only one published study of the microbiome in schizophrenia. Yolken and colleagues examined the oropharyngeal microbiome in people with schizophrenia, and found that there were increased levels of the bacteriophage, Lactobacillus phage phiadh, genome in the schizophrenia group, which were correlated with co-occurring immunological disorders (Yolken et al, 2015). There is one published study of gut microbiota in schizophrenia. Shen and colleagues found a significant reduction in butyrate producers in people with schizophrenia compared to healthy controls (Shen et al. Schiz Res, https://doi.org/10.1016/j.schres.2018.01.002).

The purpose of this study is to examine changes in serum butyrate levels with the prebiotic: Prebiotin (12g/day), an oligofructose-enriched inulin (OEI); the effect of OEI on the composition of the gastrointestinal microbiota in people with schizophrenia; and the relationship of the composition of the gut microbiota to various clinical, cognitive, and neuroimaging variables.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV-TR /DSM 5 diagnosis of schizophrenia or schizoaffective disorder;
2. Age 18-60 years
3. Clinically stable as determined by opinion of treating clinician
4. Currently treated with an antipsychotic, with no dose changes in last 14 days
5. Ability to participate in the informed consent process, as determined by a score of 10 or greater on the Evaluation to Sign Consent.
6. BMI ≤ 35

Exclusion Criteria:

1. Gastrointestinal disorders, including, but not limited to Crohn's Disease, Irritable Bowel Syndrome, Celiac Disease, whose pathology or treatment could alter the presentation or treatment of schizophrenia or significantly increase the risk associated with the proposed treatment protocol
2. Organic brain disorder, including cerebrovascular accident; epilepsy; traumatic brain injury, Loss of consciousness (LOC) for more than 30 minutes
3. Intellectual disability
4. Antibiotic or immune therapy within the last three months
5. Prebiotic or probiotic treatment within the last three months
6. Inability to understand English
7. Inability to cooperate with study procedures
8. Pregnant or lactating women secondary to pregnancy
9. Meet DSM-5 criteria for alcohol or substance use disorders (except Tobacco Use Disorder) within last 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Psychiatric Research Center (MPRC) Treatment Research Program (TRP), Catonsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buchanan RW, Werkheiser AE, Michel H, Zaranski J, Glassman M, Adams HA, Vyas G, Blatt F, Pilli NR, Pan Y, Chen S, Fraser CM, Kelly DL, Kane MA. Prebiotic Treatment in People With Schizophrenia. J Clin Psychopharmacol. 2024 Sep-Oct 01;44(5):457-461. doi: 10.1097/JCP.0000000000001899. Epub 2024 Aug 16. PMID 39146178

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four (4) participants were excluded/withdrawn prior to the initiation of study medication: one participant was excluded due to their BMI being greater than 35; one participant was excluded due to starting on an antibiotic; one participant was withdrawn because we were unable to obtain a baseline butyrate level; and one participant was discharged from the inpatient unit.
Period: Overall Study
Arm/Group | Prebiotin | Placebo
Started | 9 | 13
Completed | 8 | 12
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prebiotin | Placebo | Total
Number analyzed (Participants) | 9 | 13 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 13 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 0 | 4 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 13 | 22
Pre-Treatment Baseline Butyrate Level [Mean (Standard Deviation); unit: mg/ml] | 2.42 (0.52) | 2.34 (0.77) | 2.37 (0.67)

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Butyrate Levels
Description: We will use the following procedure to assess the effect of Prebiotin (OEI) on serum butyrate levels: there will be two test days: a) baseline (Day 0), prior to randomization to OEI or placebo; and b) Day 11, following the 10 day course of OEI/placebo treatment. We will use OEI for the inulin challenge. On the night prior to each test day, participants will receive a digestable and non-fermentable meal, e.g. lasagna. They will then fast from midnight until the morning, when they will receive their standard breakfast and OEI, 12g. We will collect fasting and 6-hour blood samples from each participant. The Day 11 change in serum butyrate levels following the OEI challenge dose (6-hour minus fasting serum butyrate level) will be compared to the Day 0 change in serum butyrate levels to determine whether the 10-day OEI treatment regimen modified the hypothesized biological signature through increased activity of butyrate-producing bacteria. Serum butyrate will be quantified by LC-MS/MS.
Time Frame: 11 days
Population: Two participants were withdrawn from the treatment phase of the study: we were unable to obtain the second challenge day butyrate levels (n=1); refusal to continue in the study (n=1).
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | Prebiotin | Placebo
Number analyzed (Participants) | 9 | 13
mg/ml
  Pre-Treatment Butyrate Level | 2.42 (0.52) | 2.34 (0.77)
  Post-Treatment Butyrate Level: number analyzed (Participants) | 8 | 12
  Post-Treatment Butyrate Level | 2.88 (1.02) | 2.40 (0.93)

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Prebiotin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/13
Other Adverse Events (participants affected / at risk) | 1/9 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prebiotin (N=9) | Placebo (N=13)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
headache (General disorders) | 0 | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT03617783/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT03617783/ICF_000.pdf